CLINICAL TRIAL: NCT01727726
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo and Active Comparator Controlled Trial of Flexible-dose Brexpiprazole (OPC-34712) as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder, the Delphinus Trial
Brief Title: A Study of Flexible-dose Brexpiprazole as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder, the Delphinus Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-12-282
Record Dates: First submitted 2012-10-31; First posted 2012-11-16 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-05

CONDITIONS: Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders
Keywords: OPC-34712; brexpiprazole; Major Depressive Disorder; Adjunctive Treatment
MeSH Terms: conditions — Depressive Disorder; Depression; Depressive Disorder, Major; Mood Disorders; Mental Disorders | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo + ADT (Placebo Comparator): Matching Placebo and assigned ADT
  Interventions: Drug: Placebo
- Brexpiprazole + ADT (Experimental): Brexpiprazole, flexible dose and assigned ADT
  Interventions: Drug: Brexpiprazole
- Seroquel XR + ADT (Active Comparator): Seroquel XR, flexible dose and assigned ADT
  Interventions: Drug: Seroquel XR

INTERVENTIONS:
Drug: Brexpiprazole — tablet/capsule
  Other Names: OPC-34712
  Arms: Brexpiprazole + ADT
Drug: Seroquel XR — tablet/capsule
  Arms: Seroquel XR + ADT
Drug: Placebo — tablet/capsule
  Arms: Placebo + ADT

SUMMARY:
To compare the efficacy of brexpiprazole (flexible dose) with placebo as adjunctive therapy to an assigned open label antidepressant therapy (ADT) in the proposed subject population with MDD.

DETAILED DESCRIPTION:
This is a trial designed to assess the safety and efficacy of brexpiprazole (flexible dose) as adjunctive therapy to an assigned known anti-depressant in depressed subjects. The trial consists of a continuous 18-week double-blind treatment period with a 30-day follow-up. Subjects who complete all trial visits through the Week 18 visit may be offered entry into an optional open-label rollover trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients 18 to 65 years of age, inclusive, at the time of informed consent.
* Subjects with both a diagnosis of MDD, and in a current major depressive episode, as defined by DSM-IV-TR criteria
* Subjects willing to discontinue all prohibited psychotropic medications to meet protocol-required washouts prior to and during the trial period.

Exclusion Criteria:

* Females who are breast-feeding and/or who have a positive pregnancy test result during screening prior to receiving trial medication
* Subject has a current Axis I (DSM-IV-TR) diagnosis of: dementia, Schizophrenia, Bipolar, Eating disorder , Obsessive-compulsive disorder, Panic disorder, Posttraumatic stress disorder
* Subjects experiencing hallucinations, delusions or any psychotic symptomatology in the current major depressive episode.
* Subjects who have met DSM-IV-TR criteria for substance abuse or dependence within the past 180 days
* Subjects currently treated with insulin for diabetes.
* Subjects with uncontrolled hypertension
* Subjects with known ischemic heart disease or history of myocardial infarction, congestive heart failure, angioplasty, stenting, or coronary artery bypass Surgery
* Subjects with a positive drug screen for cocaine, marijuana, or other illicit drugs
* Inability to swallow tablets or tolerate oral medication
* Abnormal laboratory test results, vital signs and ECG results
* Subjects who previously participated in any prior brexpiprazole clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2182 (Actual)
Dates: Start 2012-12; Primary Completion 2016-10-17 (Actual); Study Completion 2016-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hobart, Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (69):
- United States (42):
  - Birmingham, Alabama
  - Phoenix, Arizona
  - Little Rock, Arkansas
  - Bellflower, California
  - Beverly Hills, California
  - Costa Mesa, California
  - Glendale, California
  - Irvine, California
  - Redlands, California
  - San Diego, California
  - Upland, California
  - Gainesville, Florida
  - Jacksonville, Florida
  - Jacksonville Beach, Florida
  - Leesburg, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Oakland Park, Florida
  - Orange City, Florida
  - Orlando, Florida
  - Decatur, Georgia
  - Lake Charles, Louisiana
  - Baltimore, Maryland
  - Belmont, Massachusetts
  - Roslindale, Massachusetts
  - Watertown, Massachusetts
  - Creve Coeur, Missouri
  - Lebanon, New Hampshire
  - New York, New York
  - Columbus, Ohio
  - Dayton, Ohio
  - Edmond, Oklahoma
  - Portland, Oregon
  - Salem, Oregon
  - Dallas, Texas
  - Murray, Utah
  - Herndon, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Kirkland, Washington
  - Seattle, Washington
  - Brown Deer, Wisconsin
- Penticton, British Columbia, Canada
- France (6):
  - Dijon
  - Douai
  - Élancourt
  - Jarnac
  - Montepellier
  - Orvault
- Germany (4):
  - Achim
  - Mittweida
  - Stralsund
  - Würzburg
- Poland (7):
  - Bełchatów
  - Bydgoszcz
  - Gdynia
  - Kielce
  - Lublin
  - Tuszyn
  - Wroclaw
- Russia (5):
  - Arkhangelsk
  - Moscow
  - Saint Petersburg
  - Smolensk
  - Tonnelniy
- Serbia (4):
  - Belgrade
  - Kragujevac
  - Niš
  - Novi Kneževac

REFERENCES:
- [Derived] Newcomer JW, Eriksson H, Zhang P, Meehan SR, Weiss C. Changes in Metabolic Parameters and Body Weight in Patients With Major Depressive Disorder Treated With Adjunctive Brexpiprazole: Pooled Analysis of Phase 3 Clinical Studies. J Clin Psychiatry. 2019 Oct 1;80(6):18m12680. doi: 10.4088/JCP.18m12680. PMID 31577867
- [Derived] Hobart M, Zhang P, Weiss C, Meehan SR, Eriksson H. Adjunctive Brexpiprazole and Functioning in Major Depressive Disorder: A Pooled Analysis of Six Randomized Studies Using the Sheehan Disability Scale. Int J Neuropsychopharmacol. 2019 Mar 1;22(3):173-179. doi: 10.1093/ijnp/pyy095. PMID 30508090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial was conducted at 75 trial sites in 7 countries (United States, Russia, Poland, France, Serbia,Germany & Canada). Phase A non-responders entered Phase B (503 subjects randomized in 2:2:1 (197+100+206) ratio - brexpiprazole/Seroquel extended release tablets/placebo +ADT).
Pre-assignment Details: Screening period ranged from a minimum of 7 days to a maximum of 28 days and began when informed consent was signed. The purpose of the screening period was to assess eligibility criteria at 1 or more visits (as necessary to complete screening assessments) and to washout (minimum of 24 hours) prohibited concomitant pharmacotherapy, if applicable.
Groups:
- Brexpiprazole + ADT: Brexpiprazole, flexible dose and assigned ADT
  Brexpiprazole: tablet/capsule at 1 mg, 2 mg, 3 mg.
- Seroquel XR + ADT: Seroquel XR, flexible dose and assigned ADT
  Seroquel XR: tablet/capsule at 50 mg, 150 mg, 300 mg.
Period: Overall Study
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Started | 197 | 100 | 206
Completed | 171 | 86 | 186
Not Completed | 26 | 14 | 20

BASELINE CHARACTERISTICS:
Population: Randomized sample comprised all subjects who were randomized in Phase B. Subjects were considered randomized when they were assigned a treatment number by IVRS at the end of Phase A. A subject receiving IMP outside of the IVRS was not considered randomized, but safety was reported.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT | Total
Number analyzed (Participants) | 197 | 100 | 206 | 503
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 197 | 100 | 206 | 503
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (11.5) | 44.6 (11.6) | 41.8 (11.7) | 43 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 66 | 149 | 343
  Male | 69 | 34 | 57 | 160

OUTCOME MEASURES:

1. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: To determine the efficacy of brexpiprazole (flexible dose) with placebo as adjunctive therapy by assessment of MADRS total score. The MADRS depression rating scale was used to assess the subject's level of depression by utilizing the structured interview guide for the MADRS (SIGMA). The MADRS consisted of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts), each rated 0 to 6. The overall score ranged from 0 (symptoms absent) to 60 (severe depression). Lower score indicated decreased severity of depression.
Time Frame: Randomization Visit (week 8 or week 10) to End of Double-Blind Treatment (week 14 or week 16).
Population: All subjects in the Safety Sample who have an end of Phase A (ie, Week 8 or 10) value and at least one post-randomization efficacy evaluation for MADRS Total Score in Phase B.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Number analyzed (Participants) | 191 | 99 | 205
Units on a scale | -6.04 (0.43) | -4.86 (0.57) | -4.57 (0.41)
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Test type: Other; p = 0.0078, Cochran-Mantel-Haenszel; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = -1.48, 95% CI 2-sided [-2.56 to -0.39]
Statistical Analysis 2: Comparison: Seroquel XR + ADT vs Placebo + ADT; Test type: Other; p = 0.6642, Cochran-Mantel-Haenszel; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-1.63 to 1.04]

2. Secondary Outcome: Sheehan Disability Scale (SDS)
Description: To evaluate mean change in SDS score from randomization (End of Phase A) to end of Phase B. The Sheehan Disability Scale is a measurement of functional disability and impairment due to psychiatric symptoms. The SDS is a visual analogue scale that uses spatio-visual, numeric, and verbal descriptive anchors simultaneously to assess disability across the three domains ( work/social life/family life/home responsibilities). The number most representative of how much each area was disrupted by symptoms is marked along the line from 0 = not at all, to 10 = extremely. Scores of 5 and above are associated with significant functional impairment. Additionally, SDS included 2 questions related to productivity losses due to the psychiatric symptoms and impairment.
Time Frame: Randomization Visit (week 8 or week 10) to End of Double-Blind Treatment (week 14 or week 16).
Population: All subjects in the Safety Sample who have an end of Phase A (ie, Week 8 or 10) value and at least one post-randomization efficacy evaluation for SDS Score in Phase B.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Number analyzed (Participants) | 191 | 99 | 205
units on a scale | -0.97 (0.12) | -0.32 (0.16) | -0.74 (0.11)
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Test type: Other; p = 0.1334, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.52 to 0.07]
Statistical Analysis 2: Comparison: Seroquel XR + ADT vs Placebo + ADT; Test type: Other; p = 0.0237, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = 0.42, 95% CI 2-sided [0.06 to 0.78]

3. Secondary Outcome: Change From End of Phase A in MADRS Total Score for Trial Week 2 and Week 4.
Description: Change from end of Phase A in MADRS Total Score. The MADRS was used to assess the subject's level of depression by utilizing the structured interview guide for the MADRS (SIGMA). The MADRS depression rating scale was used to assess the subject's level of depression by utilizing the structured interview guide for the MADRS (SIGMA). The MADRS consisted of 10 items (apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts and suicidal thoughts), each rated 0 to 6. The overall score ranged from 0 (symptoms absent) to 60 (severe depression). Lower score indicated decreased severity of depression.
Time Frame: Change from baseline to week 2 and week 4 in Phase B (week 10/12 and week 12/14)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Number analyzed (Participants) | 191 | 99 | 205
units on a scale
  Phase B Week 2: number analyzed (Participants) | 188 | 99 | 203
  Phase B Week 2 | -2.57 (0.32) | -2.26 (0.41) | -1.04 (0.31)
  Phase B Week 4: number analyzed (Participants) | 178 | 94 | 192
  Phase B Week 4 | -4.39 (0.39) | -3.30 (0.51) | -3.22 (0.37)
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Phase B week 2; Test type: Other; p = 0.0001, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-2.29 to -0.76]
Statistical Analysis 2: Comparison: Seroquel XR + ADT vs Placebo + ADT; Phase B Week 2; Test type: Other; p = 0.0103, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = -1.22, 95% CI 2-sided [-2.15 to -0.29]
Statistical Analysis 3: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Phase B week 4; Test type: Other; p = 0.0185, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = -1.17, 95% CI 2-sided [-2.15 to -0.20]
Statistical Analysis 4: Comparison: Seroquel XR + ADT vs Placebo + ADT; Phase B Week 4; Test type: Other; p = 0.8949, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-1.27 to 1.11]

4. Secondary Outcome: Clinical Global Impression Score
Description: Mean change from end of Phase A in Clinical Global Impression - Severity of Illness scale (CGI-S) score and Improvement scale (CGI-I) during double-blind randomized Phase B treatment. CGI-S score assessed how mentally ill the patient was at that time. CGI-S score is calculated from 0 to 7 (0 indicates not assessed 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and7 indicated among the most extremely ill patient). CGI-I score is compared to his/her condition at baseline, how much has the patient changed. CGI-I score is calculated from 0 to 7 (0 indicates not assessed and 7 indicates very much worse).
Time Frame: From randomization to Phase B week 6 (14/16 weeks after randomization).
Population: All subjects in the Safety Sample who have an end of Phase A (ie, Week 8 or 10) value and at least one post-randomization efficacy evaluation for CGI-S score and CGI-I score in Phase B.
Measure: Mean (Standard Deviation); unit: Mean score
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Number analyzed (Participants) | 191 | 99 | 205
Mean score
  CGI-Severity of Illness Scale | 3.98 (0.56) | 4.07 (0.58) | 4.02 (0.58)
  CGI-Improvement Scale Score | 2.55 (0.84) | 2.71 (0.87) | 2.74 (0.83)
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; CGI-Severity of Illness Scale Score; Test type: Other; p = 0.0350, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.15, 95% CI 2-sided [-0.29 to -0.01]
Statistical Analysis 2: Comparison: Seroquel XR + ADT vs Placebo + ADT; CGI-Severity of Illness Scale Score; Test type: Other; p = 0.5601, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.22 to 0.12]
Statistical Analysis 3: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; CGI-Improvement Scale Score; Test type: Other; p = 0.0146, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.35 to -0.04]
Statistical Analysis 4: Comparison: Seroquel XR + ADT vs Placebo + ADT; CGI-Improvement Scale Score; Test type: Other; p = 0.7127, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.23 to 0.15]

5. Secondary Outcome: MADRS Response at Week 6
Description: MADRS Response Rate, where response was defined as 50% reduction in MADRS Total Score, during double-blind randomized Phase B treatment.
Time Frame: Phase B week 6 (14/16 weeks after randomization).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Number analyzed (Participants) | 191 | 99 | 205
Participants | 20 | 8 | 14
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Phase B Week 6; Test type: Other; p = 0.2242, Cochran-Mantel-Haenszel; Ratio of response rate = 1.49, 95% CI 2-sided [0.78 to 2.84]
Statistical Analysis 2: Comparison: Seroquel XR + ADT vs Placebo + ADT; Phase B Week 6; Test type: Other; p = 0.5998, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.26, 95% CI 2-sided [0.53 to 2.98]

6. Secondary Outcome: Number of Participants With MADRS
Description: MADRS Remission Rate, where remission was defined as MADRS Total Score ≤ 10 and 50% reduction in MADRS Total Score, for every trial week visit during double-blind randomized Phase B treatment.
Time Frame: Phase B week 6 (14/16 weeks after randomization).
Population: Number of subjects in the Safety Sample who had an end of Phase A (ie, Week 8 or 10) value and at least one post randomization efficacy evaluation for MADRS Total Score in Phase B.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Number analyzed (Participants) | 191 | 99 | 205
Participants | 13 | 2 | 9
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Phase B Week 6; Test type: Other; p = 0.3321, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.52, 95% CI 2-sided [0.66 to 3.49]
Statistical Analysis 2: Comparison: Seroquel XR + ADT vs Placebo + ADT; Phase B Week 6; Test type: Other; p = 0.3917, Cochran-Mantel-Haenszel; Ratio of Response Rate = 0.51, 95% CI 2-sided [0.11 to 2.46]

7. Secondary Outcome: CGI-I Response Rate
Description: CGI-I Response rate, where response was defined as a CGI-I score of 1 or 2 (very much improved or much improved), during double-blind randomized Phase B treatment.
Time Frame: Phase B week 6 (14/16 weeks after randomization).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Number analyzed (Participants) | 191 | 99 | 205
Participants | 100 | 48 | 79
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Phase B Week 6; Test type: Other; p = 0.0032, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.35, 95% CI 2-sided [1.10 to 1.66]
Statistical Analysis 2: Comparison: Seroquel XR + ADT vs Placebo + ADT; Phase B Week 6; Test type: Other; p = 0.0898, Cochran-Mantel-Haenszel; Ratio of Response Rate = 1.24, 95% CI 2-sided [0.98 to 1.59]

8. Secondary Outcome: Number of Participants With Adverse Events
Description: To evaluate the safety and tolerability of brexpiprazole (flexible dose) as adjunctive therapy to ADT in the proposed subject population with MDD as AE variables.
Time Frame: From screening (Day -28 to Day-1) upto post treatment follow-up.
Population: Randomized subjects in Phase B who received at least one dose of double-blind trial medication as indicated on the dosing record.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Number analyzed (Participants) | 197 | 100 | 206
Participants
  Death | 0 | 0 | 0
  Serious TEAE | 0 | 1 | 1
  Discontinuation due to TEAE | 2 | 4 | 1
  Any TEAE | 100 | 58 | 107

9. Secondary Outcome: Sheehan Disability Scale (SDS) Individual Item Scores.
Description: To evaluate mean change in SDS score from randomization (End of Phase A) to end of Phase B. The Sheehan Disability Scale (a self rated questionnaire) was used for measurement of functional disability and impairment due to psychiatric symptoms. The SDS is a visual analogue scale that uses spatio-visual, numeric, and verbal descriptive anchors simultaneously to assess disability across the three domains (work/school work, social life/leisure activities and family life/home responsibilities). All domains were rated on a score scale ranged from 0 (no impairment) to 10 (most severe). Score of 5 and above indicated significant functional impairment. A total score was addition of the 3 individual scores and the total score ranged from 0 (no impairment) to 30 (most severe).
Time Frame: Randomization Visit (week 8 or week 10) to End of Double-Blind Treatment (week 14 or week 16).
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
Number analyzed (Participants) | 191 | 99 | 205
units on a scale
  Work/School Score: number analyzed (Participants) | 125 | 67 | 136
  Work/School Score | -0.59 (0.16) | -0.22 (0.21) | -0.74 (0.16)
  Social Life Score | -1.03 (0.13) | -0.26 (0.17) | -0.70 (0.12)
  Family Life Score | -1.02 (0.13) | -0.34 (0.18) | -0.67 (0.13)
Statistical Analysis 1: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Work/School Score; Test type: Other; p = 0.4480, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = 0.16, 95% CI 2-sided [-0.25 to 0.56]
Statistical Analysis 2: Comparison: Seroquel XR + ADT vs Placebo + ADT; Work/School Score; Test type: Other; p = 0.0380, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = 0.52, 95% CI 2-sided [0.03 to 1.02]
Statistical Analysis 3: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Social Life Score; Test type: Other; p = 0.0436, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-0.66 to -0.01]
Statistical Analysis 4: Comparison: Seroquel XR + ADT vs Placebo + ADT; Social Life Score; Test type: Other; p = 0.0350, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = 0.43, 95% CI 2-sided [0.03 to 0.84]
Statistical Analysis 5: Comparison: Brexpiprazole + ADT vs Seroquel XR + ADT; Family Life Score; Test type: Other; p = 0.0424, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = -0.35, 95% CI 2-sided [-0.69 to -0.01]
Statistical Analysis 6: Comparison: Seroquel XR + ADT vs Placebo + ADT; Family Life Score; Test type: Other; p = 0.1230, MMRM; Mixed-model repeated measures (MMRM); Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.09 to 0.75]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from screening (Day -28 to Day-1) upto post treatment follow-up.
Description: All adverse events which started after start of double blind study drug treatment; or if the event was continuous from end of phase A and was worsening, serious, study drug related, or resulted in death, discontinuation, interruption or reduction of study therapy. Subjects in Phase B who received at least one dose of double-blind IMP as indicated on the dosing record. If a subject was dispensed IMP and was lost to follow up, he/she was considered exposed.
Arm/Group | Brexpiprazole + ADT | Seroquel XR + ADT | Placebo + ADT
All-Cause Mortality (participants affected / at risk) | 0/197 | 0/100 | 0/206
Serious Adverse Events (participants affected / at risk) | 0/197 | 1/100 | 1/206
Other Adverse Events (participants affected / at risk) | 62/197 | 33/100 | 39/206
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brexpiprazole + ADT (N=197) | Seroquel XR + ADT (N=100) | Placebo + ADT (N=206)
malignanat melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brexpiprazole + ADT (N=197) | Seroquel XR + ADT (N=100) | Placebo + ADT (N=206)
Asthenia (General disorders) | 4 | 2 | 0
fatigue (General disorders) | 3 | 4 | 3
Nasopharyngitis (Infections and infestations) | 9 | 2 | 9
Weight Increased (Investigations) | 7 | 4 | 4
Increased Appetite (Metabolism and nutrition disorders) | 5 | 5 | 2
Akathisia (Nervous system disorders) | 12 | 3 | 4
Dizziness (Nervous system disorders) | 7 | 3 | 5
Headache (Nervous system disorders) | 11 | 1 | 10
Somnolence (Nervous system disorders) | 11 | 18 | 2
Insomnia (Psychiatric disorders) | 5 | 3 | 4
Irritability (Psychiatric disorders) | 4 | 1 | 3
Restlessness (Psychiatric disorders) | 5 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes